CLINICAL TRIAL: NCT03043482
Title: A Phase 1, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of VS 105 Following Oral Administration in Healthy and Hemodialysis Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of VS 105
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vidasym, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VS 105 SAD MAD 001
Record Dates: First submitted 2017-01-27; First posted 2017-02-06 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Chronic-kidney Disease Stage 5D on Stable Hemodialysis
Keywords: VS-105; Renal Insufficiency, Chronic; Secondary hyperparathyroidism
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single VS-105/placebo to healthy (Experimental): Single ascending dose VS-105 or placebo to healthy subjects
  Interventions: Drug: Single VS-105/placebo to healthy
- Multiple VS-105/placebo to healthy (Experimental): Multiple ascending dose VS-105 or placebo to healthy subjects
  Interventions: Drug: Multiple VS-105/placebo to healthy
- Multiple VS-105/placebo to HD subjects (Experimental): Multiple ascending dose VS-105 or placebo to hemodialysis (HD) subjects
  Interventions: Drug: Multiple VS-105/placebo to HD subjects

INTERVENTIONS:
Drug: Single VS-105/placebo to healthy — In Part 1, single ascending doses of VS-105 or placebo will be administered to approximately 5 cohorts of 8 healthy subjects in each cohort with 6 receiving active and 2 receiving placebo.
  Other Names: CK15
  Arms: Single VS-105/placebo to healthy
Drug: Multiple VS-105/placebo to healthy — In Part 2, multiple ascending doses of VS 105 or placebo will be administered each morning over 7 consecutive days to approximately 3 cohorts of 8 healthy subjects in each cohort with 6 receiving active and 2 receiving placebo..
  Other Names: CK15
  Arms: Multiple VS-105/placebo to healthy
Drug: Multiple VS-105/placebo to HD subjects — In Part 3, multiple ascending doses of VS 105 will be administered over 14 consecutive days to approximately 3 cohorts that will each include 4 hemodialysis subjects with 3 receiving active drug and 1 receiving placebo.
  Other Names: CK15
  Arms: Multiple VS-105/placebo to HD subjects

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and PK following single and multiple ascending dose administration of VS-105 in healthy subjects and patients with chronic kidney disease stage 5D (CKD-5D) on hemodialysis.

DETAILED DESCRIPTION:
This is a first in human, 3 part, single and multiple ascending dose study in healthy subjects and subjects with end stage renal disease (ESRD) requiring hemodialysis (HD). A Safety Monitoring Committee (SMC) will evaluate safety data from each dose cohort before proceeding with the subsequent cohort. The SMC will also review data from each Part of the study before proceeding to the next scheduled Part.

In Part 1, single ascending doses (SAD) of VS 105 will be administered to approximately 5 dose cohorts of 8 healthy subjects each. In Part 2, multiple ascending doses (MAD) of VS 105 will be administered to approximately 3 dose cohorts of 8 healthy subjects each. VS 105 doses for MAD cohorts in Part 2 will be determined by the SMC and based on results from Part 1.

In Part 3, MAD of VS 105 will be administered to approximately 3 successive dose cohorts that will each include 4 subjects with ESRD requiring HD. VS 105 doses used in Part 3 will be selected by the SMC based on review of safety and/or pharmacokinetic (PK) results from Part 1 and Part 2.

Parts 1 & 2 of the study will assess the safety, tolerability, and PK of ascending doses of VS 105 to determine the dose range that is safe and well tolerated in healthy subjects.

Part 3 of the study will assess the safety, tolerability, and PK of various doses of VS 105 in subjects with ESRD requiring HD (ie, HD subjects), who represent the target population with secondary hyperparathyroidism (SHPT).

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects (Parts 1 & 2)

Eligible healthy subjects must meet all of the following criteria to quality for enrollment in this study:

1. Healthy male and female subjects between 18 and 60 years of age (inclusive). Healthy status, as determined by the investigator, will be based on medical and surgical history, as well as a complete physical examination including vital signs, electrocardiogram (ECG), and laboratory test results.
2. A body mass index (BMI) between 18 and 35 kg/m2 (inclusive).
3. Female subjects of childbearing potential must be non pregnant and non lactating, and have a negative serum pregnancy test at Screening and a negative serum or urine pregnancy test on Day 1 (if initial serum human chorionic gonadotropin [hCG] test results are indeterminate, follow up testing should be performed). Female subjects of childbearing potential (including perimenopausal women who have had menstrual bleeding within 1 year) must be using a method of birth control considered to be appropriate by the investigator (eg, abstinence, double barrier methods, hormonal contraceptives, or partner with vasectomy) for the entire duration of the trial. Female subjects of childbearing potential must agree to use appropriate birth control from the time of Screening until at least 1 month after their last dose of study drug.

   Women are considered to be not of childbearing potential if they are postmenopausal (defined as amenorrheic for ≥12 months with a confirmed follicle stimulating hormone [FSH] ≥ 40 mIU/mL) or if they have been surgically sterilized.
4. Male subjects must either: remain abstinent from intercourse, be sterile, or agree to use a method of birth control considered to be appropriate by the investigator (eg, condom with spermicide) from the time of Screening until 1 month after their last dose of study drug.
5. Non smoker (and no use of other tobacco or nicotine containing products) as documented by history (no nicotine use over the past 6 months) and a negative cotinine test at Screening and Day 1.
6. Capable of understanding the written informed consent form (ICF) and providing signed and witnessed written informed consent, as well as willing and able to comply with protocol requirements.

Hemodialysis Subjects (Part 3)

Eligible subjects with ESRD requiring HD must meet all of the following criteria to qualify for enrollment in this study:

1. Subject has end stage renal disease and is on a stable (defined as Kt/V ≥ 1.2 on two occasions within 3 months of screening) HD regimen (prescribed at least 3 times/week) for at least 3 months prior to screening.
2. 18 to 75 years of age (inclusive).
3. Serum calcium: 8.0 to 10.0 mg/dL; serum phosphorus: 3.0 to 7.0 mg/dL; and serum iPTH: 200 to 1000 pg/mL (at the time of Screening).
4. Subjects who have been receiving other vitamin D receptor analogs (eg, calcitriol, paricalcitol [Zemplar], doxercalciferol [Hectorol]) must allow for a washout period of 3 weeks prior to study drug administration on Day 1.

   Note: (1) If washout of VDRA therapy and/or cinacalcet is required, a check in visit should be performed 1 week into the washout period to monitor for safety (at a minimum, this visit will include laboratory testing for albumin corrected calcium; additional assessments may be performed at the investigator's discretion). (2) The 3 week duration of washout may be adjusted on a case by case basis following discussion and mutual agreement between the investigator and medical monitor.
5. A BMI between 18 and 40 kg/m2 (inclusive).
6. Female subjects of childbearing potential must be non pregnant and non lactating, and have a negative serum pregnancy test at Screening and Day 1 (if initial serum hCG test results are indeterminate, follow up testing should be performed). Female subjects of childbearing potential (including perimenopausal women who have had menstrual bleeding within 1 year) must be using a method of birth control considered to be appropriate by the investigator (eg, abstinence, double barrier methods, hormonal contraceptives, or partner with vasectomy) for the entire duration of the trial. Female subjects of childbearing potential must agree to use appropriate birth control from the time of Screening until 1 month after their last dose of study drug.

   Women are considered to be not of childbearing potential if they are postmenopausal (defined as amenorrheic for ≥12 months with a confirmed FSH ≥ 40 mIU/mL) or if they have been surgically sterilized.
7. Male subjects must either: remain abstinent from intercourse, be sterile, or agree to use a method of birth control considered to be appropriate by the investigator (eg, condom with spermicide) from the time of Screening until 1 month after their last dose of study drug.
8. Capable of understanding the written ICF and providing signed and witnessed written informed consent, as well as willing and able to comply with protocol requirements.
9. Considered to be clinically stable with respect to underlying renal impairment, as determined by investigator, and based upon a medical evaluation that includes a medical history, physical examination, laboratory tests and ECG.
10. Subjects who need concurrent medications must have a medication regimen considered to be stable by the investigator (eg, no new drugs or significant changes to dosage[s] within 14 days prior to study drug administration on Day 1; no changes expected during study conduct). Changes of medications in HD subjects are subject to dialysis site protocols such that erythropoiesis stimulating agents (ESAs) and iron can be changed based on the current subject status, the dialysis unit's standard of practice, and subject safety. Changes to medications may be allowed at the discretion of the investigator.
11. Subjects must have satisfactory control of blood pressure (as determined by the investigator), and blood pressure at Screening must be ≤ 140/90 mmHg with confirmatory repeat measurements allowed per the CRU's standard operating procedures (SOPs).

Exclusion criteria:

Hemodialysis Subjects (Part 3)

Subjects undergoing hemodialysis who meet any of the following criteria will be excluded from the study:

1. Receiving blood purification therapy other than hemodialysis.
2. Dialysis via central venous catheter.
3. Expected to undergo pre emptive or scheduled renal transplant within 6 months after Screening.
4. Pregnant (positive pregnancy test) or lactating women, and male subjects whose female partners are pregnant or lactating. If serum hCG pregnancy test results are indeterminate, follow up testing should be performed to determine eligibility.
5. History of significant gastrointestinal, hepatic, broncho pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis, or any other unstable or new onset medical conditions that, in the opinion of the investigator, would constitute a risk factor for study participation or receipt of study drug.
6. ECG heart rate (HR) <45 bpm or HR >100 bpm; QTcF >500 ms.
7. History of having received or currently receiving any systemic anti neoplastic (including radiation) or immune modulatory treatment (including systemic oral corticosteroids) ≤ 6 months prior to the first dose of study drug or such treatment is expected to be needed at any time during the study.
8. Subjects who have had significant acute infection (eg, influenza, local infection, acute gastrointestinal symptoms) or any other clinically significant illness within 2 weeks prior to the first dose of study drug.
9. History of significant gastrointestinal diseases (such as gastric or duodenal ulcers) that affect the absorption of the study drug. Subjects with a history of gastrointestinal disease may be allowed if there is no evidence of active disease for 3 months prior to Day 1 or at the discretion of the investigator.
10. Any confirmed significant allergic reactions (anaphylaxis or angioedema) against any drug, or multiple drug allergies (non active hay fever is allowable per the investigator's discretion).
11. Any clinically significant concomitant disease or condition (including treatment for such conditions) that could either interfere with or, in the opinion of the investigator, pose an unacceptable risk to the subject.
12. Positive test at Screening for Hepatitis B (HBsAg) or human immunodeficiency virus (HIV Ab). If a subject has positive test results for Hepatitis C (HCV RNA or HCVAb) but liver function tests are otherwise not clinically significant, the subject may be included at the investigator's discretion.
13. Any other clinically significant abnormalities in laboratory test results at Screening. In the case of uncertain or questionable results, tests performed during Screening may be repeated before the first dose of study drug to confirm eligibility.
14. Treatment with another investigational drug or device study within 30 days or 5 half lives (whichever is longer) prior to Screening.
15. Positive test for drugs of abuse and/or positive alcohol test at Screening or Day 1.
16. History of drug abuse or addiction within 6 months prior to Screening.
17. History (within 3 months of Screening) of alcohol consumption exceeding an average of 2 standard drinks per day (1 standard drink = 10 grams of alcohol). Alcohol consumption will be prohibited, at a minimum, within 48 hours before Screening, and from 48 hours before until 48 hours after each dose, and within 48 hours before each scheduled visit.
18. Use of > 5 cigarettes (or equivalent nicotine containing product) per day.
19. Use of the following:

    1. any prescribed medications or herbal remedies within 3 weeks prior to first dosing, including any prescribed vitamin D analogs, cinacalcet, phosphate binders, and other agents that affect serum calcium and iPTH levels. Exceptions may be made at the discretion of the investigator including subjects on a stable dose of calcimimetics and/or phosphate binders for 3 months prior to first dosing;
    2. use of any OTC medications (including vitamins and supplements) within 2 weeks prior to first dosing, unless specifically indicated for an underlying concomitant condition.

    Note: exceptions may be made to this criterion (#19) on a case by case basis following discussion and agreement between the investigator and the medical monitor.
20. Planned parathyroid intervention during the study period.
21. Use of medications or nutrients known to modulate CYP3A and/or 5' diphospho glucoronosyltransferase (UGT) activity, based on the VS 105 metabolic pathway:

    1. strong or moderate inhibitors of CYP3A4 and/or UGT within 2 weeks prior to first dose administration, including but not limited to the following drugs: ketoconazole, miconazole, itraconazole, fluconazole, atazanavir, erythromycin, clarithromycin, ranitidine, cimetidine, verapamil, and diltiazem;
    2. any strong or moderate inducer of CYP3A4 and/or UGT, within 4 weeks prior to first dose administration, including but not limited to the following drugs: rifampicin, rifabutin, glucocorticoids, carbamazepine, phenytoin, phenobarbital, and St. John's wort.

    Note: at the discretion of the investigator, the study pharmacist and/or medical monitor may review the subject's medication list to assist with eligibility determination in regard to this criterion (#21).
22. Subjects under judicial supervision, guardianship or curatorship, or with other medical or social conditions that would potentially interfere with the subject's ability to comply with the study visit schedule or the study assessments.
23. Blood donation or significant blood loss (ie, > 500 mL) within 56 days prior to Day 1.
24. Plasma or platelet donation within 14 days prior to Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple ascending doses of VS 105 administered orally to healthy and HD subjects (numbers and percentages of adverse events). | 3 weeks
  Adverse events will be counted within each treatment and study part. The numbers and percentages of adverse events will be tabulated by body system, preferred term, and severity.
Pharmacokinetic (PK) of VS-105 in serum: area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration | pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 and 16 hours and 2, 3, 7, 8, 9, 14, 15, 16 days after dosing.
  AUC0-last: The area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration.
PK of VS-105 in serum: area under the serum concentration-time curve from time zero to infinity. | pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 and 16 hours and 2, 3, 7, 8, 9, 14, 15, 16 days after dosing.
  AUC0-∞: The area under the serum concentration-time curve from time zero to infinity
PK of VS-105 in serum: observed maximum serum concentration following drug administration | pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 and 16 hours and 2, 3, 7, 8, 9, 14, 15, 16 days after dosing.
  Cmax: The observed maximum serum concentration following drug administration
PK of VS-105 in serum: terminal elimination half-life | pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 and 16 hours and 2, 3, 7, 8, 9, 14, 15, 16 days after dosing.
  T1/2: The terminal elimination half-life
PK of VS-105 in serum: time to reach the maximum concentration after drug administration | pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 and 16 hours and 2, 3, 7, 8, 9, 14, 15, 16 days after dosing.
  Tmax: The time to reach the maximum concentration after drug administration

SECONDARY OUTCOMES:
Serum calcium (ionized) in healthy and HD subjects | Pre-dose and 1, 2, 15, 21 days after dosing
  To evaluate the changes from baseline in concentrations of serum calcium (ionized) in healthy and HD subjects after multiple doses of VS 105 (Part 2 and Part 3 only).
Serum phosphorous in healthy and HD subjects | Pre-dose and 1, 2, 15, 21 days after dosing
  To evaluate the changes from baseline in concentrations of serum phosphorous in healthy and HD subjects after multiple doses of VS 105 (Part 2 and Part 3 only).
Serum intact parathyroid hormone (iPTH) in healthy and HD subjects | Pre-dose and 1, 2, 15, 21 days after dosing
  To evaluate the changes from baseline in concentrations of serum intact parathyroid hormone (iPTH) in healthy and HD subjects after multiple doses of VS 105 (Part 2 and Part 3 only).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Hardies, Study Director — Davita Clinical Research; Robert Williams, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No